CLINICAL TRIAL: NCT04785781
Title: Effects of Face Masks on Cardiopulmonary Capacity in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erhan KIZMAZ, Msc, Research Assitant, Pamukkale University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: pamukkaleU:
Record Dates: First submitted 2021-02-24; First posted 2021-03-08 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Covid-19
Keywords: covid19; cardiopulmoary; exercise capacity; face masks
MeSH Terms: conditions — COVID-19 | interventions — Masks; Long-Term Synaptic Depression

STUDY DESIGN:
Intervention Model Description: individuals will perform cycle ergometer without mask, with surgical mask and FFP2/N95. there will be 48 hours wash-out between tests.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no mask (Other): individuals perform cardiopulmonary test via cycle ergometer without mask till voluntary exhaustion
  Interventions: Other: without masks
- surgical mask (Other): individuals perform cardiopulmonary test via cycle ergometer with surgical mask till voluntary exhaustion
  Interventions: Other: Surgical face mask (Vheal Med Co., Ltd., Istanbul, Turkey)
- N95/fpp2 (Other): individuals perform cardiopulmonary test via cycle ergometer with N95 mask till voluntary exhaustion
  Interventions: Other: FFP2\N95 protective face mask (Musk protective technology, Gaziantep, Turkey)

INTERVENTIONS:
Other: without masks — apply a bicycle ergometer test protocol to individuals without a mask
  Arms: no mask
Other: Surgical face mask (Vheal Med Co., Ltd., Istanbul, Turkey) — apply a bicycle ergometer test protocol to individuals with a surgical mask
  Arms: surgical mask
Other: FFP2\N95 protective face mask (Musk protective technology, Gaziantep, Turkey) — apply a bicycle ergometer test protocol to individuals with a FFP2\N95 mask
  Arms: N95/fpp2

SUMMARY:
The aim of our study is to compare the effects of face masks on cardiopulmonary capacity in young healthy individuals. The results of our study will show the effects of face masks commonly used during the pandemic period.

DETAILED DESCRIPTION:
The aim of our study is to compare the effects of face masks on cardiopulmonary capacity in young healthy individuals. The results of our study will show the effects of face masks commonly used during the pandemic period.

The hypotheses we will test for this purpose; H1: face masks affect cardiopulmory capacity in healthy individuals H2: face masks affect heart rate in health individuals H3: face masks affect oxygen saturation in healthy individuals H4: face masks affect respiratory frequency in healthy individuals

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to 30
* healthy young individuals

Exclusion Criteria:

* having cardiovasculary conditions
* having respiratory conditions
* having inflammatory conditions
* any contraindicated situations for cardiopulmonary tests

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
time to exhaustion | 5-10 minutes
  individuals perform cardiopulmonary capacity test with cycle ergometer till voluntary exhaustion
Mask comfort/discomfort | 5-10 minutes
  Mask comfort/discomfort will be assesed by published questionnaire quantify the following ten domains of comfort/discomfort of wearing a mask: humidity, heat, breathing resistance, itchiness, tightness, saltiness, feeling unfit, odor, fatigue, and overall discomfort

SECONDARY OUTCOMES:
heart rate | 1 minute
  heart rate before and after test
oxygen saturation | 1 minute
  oxygen saturation via pulse oximeter before and after test
respiratory frequency | 1 minute
  Respiratory rate measured within 1 minute before and after the test

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ünver, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No